CLINICAL TRIAL: NCT00526487
Title: Evaluation of the Safety and Effectiveness Performance of the Zenith® Dissection Endovascular System in the Treatment of Patients With Aortic Dissection Involving the Descending Thoracic Aorta
Brief Title: Clinical Study to Assess Safety and Effectiveness of the Zenith® Dissection Endovascular System in Patients With Aortic Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Cook Europe (Industry)
Collaborators: Cook Group Incorporated (Industry); MED Institute, Incorporated (Industry); William Cook Australia (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 07-004; 370010, TXD
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Aortic Dissection Involving the Descending Thoracic Aorta
Keywords: Thoracic Dissection; Dissection; Endovascular
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Endovascular Repair
  Interventions: Device: Zenith® Dissection Endovascular System; Device: Endovascular Repair

INTERVENTIONS:
Device: Zenith® Dissection Endovascular System — The Zenith® Thoracic Dissection Study is a clinical trial to study the safety and effectiveness of the Zenith® Dissection Endovascular System in the treatment of dissections (length-wise tear) of the descending thoracic aorta. The Zenith® Dissection Endovascular System is comprised of the Zenith TX2® TAA Endovascular Graft and the Zenith® Dissection Endovascular Stent. Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the graft and the dissection stent into place in the aorta.
Device: Endovascular Repair — Endovascular Repair

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness performance of the Zenith® Dissection Endovascular System in the treatment of aortic dissections involving the descending thoracic aorta.

DETAILED DESCRIPTION:
The Zenith® Thoracic Dissection Study is a clinical trial to study the safety and effectiveness of the Zenith® Dissection Endovascular System in the treatment of dissections (length-wise tear) of the descending thoracic aorta. The Zenith® Dissection Endovascular System is comprised of the Zenith TX2® TAA Endovascular Graft and the Zenith® Dissection Endovascular Stent. Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the graft and the dissection stent into place in the aorta.

ELIGIBILITY:
Inclusion Criteria:

* Branch vessel obstruction/compromise
* Peri-aortic effusion/hematoma
* Resistant hypertension
* Persistent pain/symptoms
* Transaortic growth greater than or equal to 5 mm within 3 months (or transaortic diameter greater than or equal to 40 mm)

Exclusion Criteria:

* Age less than 18 years
* Frank rupture
* Diagnosed or suspected congenital degenerative connective tissue disease
* Systemic infection
* Untreatable reaction to contrast
* Surgical/endovascular AAA repair within 30 days
* Previous placement of thoracic endovascular graft
* Prior repair of descending thoracic aorta
* Interventional/open procedures within 30 days
* Onset of symptoms > 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is survival at 30 days | 30 days

SECONDARY OUTCOMES:
Measure: Clinical utility, incidence and rate of adverse events, mortality, factors related to morbidity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lombardi, MD, Principal Investigator — Thomas Jefferson University
Locations (8):
- St. Vincent's Hospital Melbourne, Melbourne, Australia
- St. Anne's Universtiy Hospital Brno, Brno, Czechia
- CHRU de Lille, Lille, Cedex, France
- Germany (3):
  - Hannover Medical School, Hanover
  - Heart Center Leipzig / Park Hospital, Leipzig
  - Clinic of Internal Medicine, University Hospital Rostock, Rostock
- Italy (2):
  - Hospital San Raffaele, Milan
  - IRCCS Policlinico San Matteo, Pavia

REFERENCES:
- [Derived] Lombardi JV, Cambria RP, Nienaber CA, Chiesa R, Mossop P, Haulon S, Zhou Q; STABLE I Investigators. Five-year results from the Study of Thoracic Aortic Type B Dissection Using Endoluminal Repair (STABLE I) study of endovascular treatment of complicated type B aortic dissection using a composite device design. J Vasc Surg. 2019 Oct;70(4):1072-1081.e2. doi: 10.1016/j.jvs.2019.01.089. Epub 2019 May 28. PMID 31147139